CLINICAL TRIAL: NCT04092829
Title: Impact of Corpus Luteum Presence or Absence in the Incidence of Preeclampsia After Frozen Embryo Transfer
Acronym: PREECLAM-2019
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: under-recruitment
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Collaborators: IVI Bilbao (Other); IVI Barcelona (Other); IVI Madrid (Other); Vida Recoletas Sevilla (Other); IVI Vigo (Other); IVI Roma (Other); Hospital Universitario La Paz (Other); IVI Mallorca (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1906-VLC-067-JB
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Pre-Eclampsia; Frozen Embryo Transfer
Keywords: Pre-Eclampsia; Corpus Luteum; Frozen embryo transfer; Endometrial preparation
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Intervention Model Description: Randomized prospective analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FROZEN EMBRYO TRANSFER IN NATURAL CYCLE (No Intervention): After confirming ovarian rest (follicles < 10 mm) with menstruation by means of vaginal ultrasound, an ultrasound control of the natural cycle will be carried out, inducing ovulation when an ovulatory follicle of size ≥ 17mm and an endometrium ≥ 7mm are found. Serum estradiol and progesterone values will be determined that day. This induction will be carried out with an ampoule of 250 μg of rHCG (Ovitrelle®). After the injection of Ovitrelle®, the administration of micronized vaginal progesterone (Progeffik® or Utrogestan®) 200 mg/ 12 hours and 7 days after the injection, thawing and transfer of a frozen euploid blastocyst will begin 48 hours later.
- FROZEN EMBRYO TRANSFER IN SUBSTITUTED CYCLE (Active Comparator): After confirming ovarian rest (follicles < 10 mm) with menstruation by vaginal ultrasound, hormone replacement therapy with oestrogens (6 mg/day of oral oestradiol valerate - Progynova® or Progyluton®- or 150 ug/48 h of oestradiol in patches - Evopad®) will be started on day 2-3 of the cycle. On day 10-15 of treatment an ultrasound scan will be performed to assess endometrial growth and ovarian rest. After confirming an endometrial thickness ≥ 7mm by vaginal ultrasound, ovaries with follicles smaller than 10 mm, blood estradiol >100 pg/ml and serum progesterone < 1 ng/ml, luteal phase support will begin with the administration of 400 mg of micronized vaginal progesterone every 12 hours, a total of 10 shots, prior to embryo transfer of a thawed euploid blastocyst. same day. If the level of serum progesterone on the day of transfer is less than 9.2 ng/ml, a daily injection of subcutaneous progesterone (Prolutex®) will be added on the same day.
  Interventions: Procedure: FROZEN EMBRYO TRANSFER IN SUBSTITUTED CYCLE

INTERVENTIONS:
Procedure: FROZEN EMBRYO TRANSFER IN SUBSTITUTED CYCLE — The intervention group will be prepared with hormone replacement therapy with estrogens according to usual clinical practice. Frozen embryos will be transferred after ten doses of exogenous progesterone.
  Arms: FROZEN EMBRYO TRANSFER IN SUBSTITUTED CYCLE

SUMMARY:
Identifying modifiable factors that contribute to preeclampsia risk associated with assisted reproduction can improve maternal health. Recent studies have shown an increased risk for hypertensive disorders of pregnancy after in vitro fertilization, particularly for pregnancies occurring during a hormone replacement therapy such a donor egg recipient and a frozen embryo transfer. This risk may be partly attributable to the degree by which the assisted reproductive treatment affects the maternal hormonal environment, when the corpus luteum is a major source of reproductive hormones. On the other hand, cryopreserved embryos are usually thawed and replaced in in a natural or hormonally manipulated cycle; on this point, frozen embryo transfer is associated with better perinatal outcome regarding preterm birth and low birth weight yet higher risk of large for gestational age and macrosomia compared to fresh transfer. The objective of our study is to investigate whether the absence of corpus luteum adversely affects pregnancy and to analyse if there are differences in the perinatal outcomes due to differences in the endometrial preparation protocol for a frozen embryo transfer.

ELIGIBILITY:
Inclusion criteria

* All patients who, after IVF-PGT-A treatment with their own oocytes, present a euploid embryo for transfer.
* Transfer of a single euploid embryo

Exclusion criteria:

* Moderate or high smoking (> 5 cigarettes/day)
* BMI ≥30 kg/m2
* Chronic hypertension
* History of preeclampsia in previous pregnancies
* History of delayed uterine growth and placental insufficiency in previous pregnancies
* Use of donor sperm
* Woman's age ≥44 years
* Women with menstrual cycles longer than 35 days

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 591 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of pre-eclampsia during pregnancy. | 12 months
  Presence or absence of pre-eclampsia during pregnancy

SECONDARY OUTCOMES:
Bleeding during pregnancy | 12 months
  Presence or absence of Bleeding during pregnancy
Hypertension during pregnancy | 12 months
  Presence or absence of Hypertension during pregnancy
Eclampsia during pregnancy | 12 months
  Presence or absence of Eclampsia during pregnancy
Preeclampsia during pregnancy | 12 months
  Presence or absence of Preeclampsia during pregnancy
Retarded intrauterine growth during pregnancy | 12 months
  Presence or absence of retarded intrauterine growth at birth
Premature detachment of normoinserted placenta during pregnancy | 12 months
  Presence or absence of premature detachment of normoinserted placenta during pregnancy
Type II Diabetes during pregnancy | 12 months
  Presence or absence of Type II Diabetes during pregnancy
Help Sindrome during pregnancy | 12 months
  Presence or absence of Help Sindrome during pregnancy
Alterations in the volume of the amniotic fluid during pregnancy | 12 months
  Presence or absence of alterations in the volume of the amniotic fluid during pregnancy
Preterm premature rupture of membranes during pregnancy. | 12 months
  Presence or absence of preterm premature rupture of membranes during pregnancy
Fetal death | 12 months
  Presence or absence of fetal death at birth.

CONTACTS AND LOCATIONS:
Overall Officials: JOSE BELLVER PRADAS, MDPhD, Principal Investigator — IVIRMA VALENCIA
Locations (1):
- Ivi Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided